CLINICAL TRIAL: NCT06300476
Title: Safety and Efficacy of a Single Subretinal Injection of JWK006 Gene Therapy in Subjects With Stargardt Disease(STGD1)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Fang Lu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1511
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Stargardt Disease 1
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): Subretinal injection low dose of JWK006 in one eye
  Interventions: Genetic: JWK006
- Medium dose group (Experimental): Subretinal injection medium dose of JWK006 in one eye
  Interventions: Genetic: JWK006
- High dose group (Experimental): Subretinal injection high dose of JWK006 in one eye
  Interventions: Genetic: JWK006

INTERVENTIONS:
Genetic: JWK006 — Subretinal administration of gene therapy vector JWK006 to one eye.

SUMMARY:
The purpose of the study is to assess the safety and efficacy of JWK006 in Stargardt Disease(STGD1).

JWK006 is packed by adeno-associated virus vector that expressing ABCA4 gene.

DETAILED DESCRIPTION:
This clinical study is a single-center, non-randomized, non-blinded, self-controlled, dose-escalation clinical study, aiming to evaluate the safety, tolerability, and preliminary effectiveness of JWK006 injection in the treatment of approximately 12 patients(aged 10 to 18 years) with Stargardt Disease(STGD1),genotyped with ABCA4 gene mutations.

In this study, a "3+3" dose escalation trial was adopted, with 3 doses (low dose, medium dose, and high dose) set up, and 9 subjects were planned to be enrolled, 3 in each dose group. Following the principle of dose escalation, starting from the low-dose treatment group, one subject was enrolled in each dose group. In order to fully protect the safety of subjects, it is required to adopt an orderly enrollment method within each dose group, with one subject enrolled at a time. No obvious toxic or side effects are observed 28 days after the completion of the administration. The next subject in the group. At the same time, 28 days after the last subject in each dose group is administered, the researchers and others will jointly evaluate the safety results of the dose group before deciding whether to enter the next dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the informed consent form (underage subjects must be signed by their guardians), and be able to cooperate with the tests required in various studies according to the protocol requirements;
2. Aged 10 to 18 years old (including the critical value, subject to the time of signing the informed consent form), regardless of gender;
3. Clinical diagnosis of Stargardt disease(STGD1), macular changes consistent with the clinical manifestations of Stargardt disease(STGD1);
4. The biallelic ABCA4 pathogenic mutation has been confirmed by genetic testing and does not carry other pathogenic mutations for ophthalmic genetic diseases;
5. The best corrected visual acuity of the study eye is ≤ETDRS 68 letters (20/50); the best corrected visual acuity of the fellow eye is ≥20/400.

Exclusion Criteria:

1) The study eye has other conditions that may cause vision loss (such as optic atrophy, advanced glaucoma, and uveitis); (2) The presence of lens, cornea or other refractive stromal opacity in the study eye affects retinal observation and examination; (3) There are eye conditions that affect subretinal injection, or eye conditions that affect the judgment of the study endpoint; (4) Those who have undergone intraocular surgery in the study eye within 6 months; (5) Patients with AAV8 neutralizing antibody titer ≥1:1000; (6) Have received any gene therapy or cell therapy in the past; (7) Subjects of childbearing age are unwilling to use contraceptive measures; (8) One of the following situations exists: the researcher believes that there is an active infection that may affect the patient's participation in the study or that affects the study results and requires systemic treatment; hepatitis B surface antigen is positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) copies number > ULN; hepatitis C virus (HCV) antibody positive, and HCV-RNA copy number > ULN; Treponema pallidum antibody positive; human immunodeficiency virus (HIV) antibody positive; (9) Malignant tumors diagnosed within 5 years before screening (except for adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer, and breast ductal carcinoma in situ after radical mastectomy); (10) Suffering or having suffered from systemic immune system diseases; (11) Abnormal laboratory values considered to be clinically significant: alanine aminotransferase and/or aspartate aminotransferase >2.5×ULN, total bilirubin >1.5×ULN, serum creatinine >1.5×ULN, prothrombin time ≥1.5× ULN, activated partial thromboplastin time ≥1.5×ULN; (12) There is severe allergy or known allergy to the drugs used for treatment or examination in the research protocol, including allergy to study drugs; (13) Pregnant and lactating women; subjects with childbearing potential who are unable to take effective contraceptive measures within 2 weeks before screening to 6 months after administration; (14) Other circumstances that the researcher believes are not suitable for participating in this study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety(Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events) | 5 years (Screening to 5 years post JWK006 administration)
  The primary outcome measures are safety, determined by the number of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Visual acuity | 5 years (Screening to 5 years post JWK006 administration)
  Visual acuity of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS)
Ophthalmoscope Measurement | 5 years (Screening to 5 years post JWK006 administration)
  Usese Slit-lamp Biomicroscopy to visualize the anatomy of ocular structures before and after sub-retinal injections and follow-up visits.
Qualitative and quantitative assessments of autofluorescence pattern (FAF) | 5 years (Screening to 5 years post JWK006 administration)
  Changes in FAF intensity will be assessed from baseline measurements to assess damage to photoreceptors and retinal pigment epithelium cells.
multifocal electroretinogram (mfERG) | 5 years (Screening to 5 years post JWK006 administration)
  mfERG can be used to assess macular function of retina.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China